CLINICAL TRIAL: NCT02806453
Title: Effect of Magnesium Alginate on Gastroesophageal Reflux in Infants.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Prof. Maria Elisabetta Baldassarre, MD, Policlinico Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ALNEO1
Record Dates: First submitted 2016-06-16; First posted 2016-06-20 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Group A (Active Comparator): Group A: Mg alginate/thickened formula
  Interventions: Dietary Supplement: thickened formula; Dietary Supplement: Mg alginate; Behavioral: reassurance with lifestyle changes
- Group B (Active Comparator): Group B: thickened formula/Mg alginate
  Interventions: Dietary Supplement: thickened formula; Dietary Supplement: Mg alginate; Behavioral: reassurance with lifestyle changes

INTERVENTIONS:
Dietary Supplement: thickened formula
Dietary Supplement: Mg alginate
Behavioral: reassurance with lifestyle changes

SUMMARY:
A randomized controlled cross-over trial in full-term infants affected by symptoms suggestive of GER, evaluated through a validated questionnaire (Infant Gastroesophageal Reflux Questionnaire Revised).

The parents of all of the enrolled infants will be reassured on the benign nature of the condition and will advise to apply lifestyle changes for one week.

Than, the patients will be randomized into one of the two sequence treatment groups. (group A: Mg alginate/thickened formula; group B: thickened formula/Mg alginate) for two weeks. Evaluation of symptom scores will be performed at day 0, day 7, day 21 and day 35.

ELIGIBILITY:
Inclusion Criteria:

* full-term ages 3 to 12 months, affected by symptoms suggestive of GER.
* infant regurgitation defined according to the Rome IV criteria
* informed consent

Exclusion Criteria:

* Evidence of chronic diseases, hepatic, renal, or cardiac diseases, metabolic or central nervous system diseases, or use of acid suppressor treatment (H2-receptor antagonists or proton pump inhibitors [PPIs]), thickened formula, or a history of prematurity or atopy

Ages: 3 Months to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 99 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of symptom scores | From day 0 to day 35
  Infant Gastroesophageal Reflux Questionnaire Revised

CONTACTS AND LOCATIONS:
Locations (1):
- Dept Of Obstetrics and Neonatology - Section of Neonatology University of Bari Policlinico Hospital, Bari, Italy